CLINICAL TRIAL: NCT04157725
Title: Mild Stimulation Protocol Using Clomiphene Citrate / Gonadotropins Versus Conventional Stimulation Protocol for Women With PCOS Undergoing in Vitro Fertilization (IVF): a Prospective Non-randomized Controlled Trial
Brief Title: Mild Stimulation Protocol Using Clomiphene Citrate for Women With PCOS Undergoing in Vitro Fertilization
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Johnny Awwad, Professor of Obstetrics and Gynecology, American University of Beirut Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AmericanUBMC-MS
Record Dates: First submitted 2019-07-17; First posted 2019-11-08 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: PCO - Polycystic Ovaries; Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (mild stimulation protocol) (Experimental)
  Interventions: Drug: mild stimulation protocol: oral Clomiphene Citrate
- Group B (conventional stimulation protocol) (Active Comparator)
  Interventions: Drug: Conventional Stimulation Protocol: will receive FSH/HMG

INTERVENTIONS:
Drug: mild stimulation protocol: oral Clomiphene Citrate — Group A (mild stimulation protocol) will receive oral Clomiphene Citrate (Clomid®) 150 mg/day for 5 days (starting on the 2nd of menses), followed by FSH/HMG (human menopausal gonadotropins) at a daily dose of 150-225 IU starting from the 6th day of the menstrual cycle. GnRH antagonist (Cetrotide®, Merck-Serono, Switzerland) 0.25 mg subcutaneously daily will be started once a dominant follicle becomes ≥14 mm until the day of final follicle maturation. Once 3 leading follicles reach 18mm in diameter, final follicle maturation will be triggered using HCG (Choriomon® 10,000 IU) in the presence of 14 or less pre-ovulatory follicles or GnRH agonist (Triptorelin-Gonapeptyl® 0.3mg single dose) in the presence of 15 or more follicles. The choice of the starting FSH/HMG daily dose will be tailored to BMI: 150 IU/d for BMI less than 25 and 225IU/d for BMI 25 and above.
  Arms: Group A (mild stimulation protocol)
Drug: Conventional Stimulation Protocol: will receive FSH/HMG — Group B (conventional stimulation protocol) will receive FSH/HMG (human menopausal gonadotropins) at a daily dose of 150-225 IU starting on the 2nd day of menses. GnRH antagonist (Cetrotide®, Merck-Serono, Switzerland) 0.25 mg subcutaneously daily will be started once a dominant follicle becomes ≥14 mm until the day of final follicle maturation. Once 3 leading follicles reach 18mm in diameter, final follicle maturation will be triggered using HCG (Choriomon® 10,000 IU) in the presence of 14 or less pre-ovulatory follicles or GnRH agonist (Triptorelin-Gonapeptyl® 0.3mg single dose) in the presence of 15 or more follicles. The choice of the starting FSH/HMG daily dose will be tailored to BMI: 150 IU/d for BMI less than 25 and 225IU/d for BMI 25 and above.
  Arms: Group B (conventional stimulation protocol)

SUMMARY:
Infertility is of increasing significance affecting almost 48.5 million couples around the world. Anovulation is a major cause of infertility in women with polycystic ovary syndrome (PCOS) accounting for about 80% of women with anovulatory infertility. Ultrasound morphological features of PCOS include the presence of 16 or more follicles measuring 2-9 mm in diameter, and/or an overall large ovarian volume of >10mm3. Women with PCOS ultrasound features exhibit an exaggerated response to controlled ovarian stimulation.

Controlled ovarian hyperstimulation is an established prerequisite to assisted reproductive techniques with the aim of obtaining a higher yield of oocytes and ultimately increasing success rates. According to the ESHRE/ASRM consensus on infertility treatment related to polycystic ovary syndrome, IVF seems to represent a reasonable treatment option as the risks of multiple pregnancies and ovarian hyper-stimulation syndrome may be kept to a minimum. The optimal stimulation protocol however is still debatable. Recently, patient-friendly stimulation protocols for assisted reproductive technology were introduced aiming at minimizing overall treatment costs and health hazards to the patient. Mild stimulation protocols are considered relatively novel protocols. They consist of combining oral stimulation agents (clomiphene citrate or letrozole) with low-dose gonadotropins as effective alternatives to conventional gonadotropin-only stimulation protocols. Mild stimulation protocol has been associated with better tolerance, ease of use, and comparable livebirth outcomes. The investigators aim to test the hypothesis that mild stimulation protocols could produce a similar proportion of term livebirths to conventional treatment, while reducing treatment costs and health hazards.

This is a prospective non-randomized controlled trial comparing a mild ovarian stimulation protocol to conventional treatment for assisted reproductive technology at the Division of Reproductive Endocrinology and Infertility - Haifa Idriss Fertility Center - American University of Beirut Medical Center.

DETAILED DESCRIPTION:
Infertility is a medical condition of increasing significance with an estimated 48.5 million affected couples around the world . Anovulation is a major cause of infertility in women with polycystic ovary syndrome (PCOS) accounting for about 80% of women with anovulatory infertility. The prevalence of PCOS varies widely among different ethnic populations and is highest in the Middle East. One way to diagnose PCOS is on the basis of the Rotterdam criteria, according to which women should satisfy 2 of 3 criteria including anovulation, polycystic ovarian morphology on ultrasound and hyperandrogenism (either clinical or biochemical). Trans-vaginal ultrasound evaluation is an important tool to assess ovarian features and determine the risk for ovarian hyper-response to follicle stimulation.

Ultrasound morphological features of polycystic ovary syndrome (PCOS) include the presence of 16 or more follicles measuring 2-9mm in diameter, and/or an overall large ovarian volume of >10mm3. Women with PCOS ultrasound features exhibit an exaggerated response to controlled ovarian stimulation . It was demonstrated that the number of baseline follicles seen on ultrasound strongly correlates with the number of recovered oocytes, and that was especially documented in women with a baseline number of pre-antral follicles exceeding 15 who were found to be at increased risk for ovarian hyper-stimulation syndrome .

Controlled ovarian hyperstimulation is an established prerequisite to assisted reproductive techniques with the aim of obtaining a higher yield of oocytes and ultimately increasing success rates. According to the ESHRE/ASRM consensus on infertility treatment related to polycystic ovary syndrome (2008), IVF seems to represent a reasonable treatment option as the risks of multiple pregnancies and ovarian hyper-stimulation syndrome may be kept to a minimum. The optimal stimulation protocol however is still debatable.

The investigators plan to conduct a prospective non-randomized controlled trial comparing a mild ovarian stimulation protocol to conventional treatment for assisted reproductive technology at the Division of Reproductive Endocrinology and Infertility - Haifa Idriss Fertility Center - American University of Beirut Medical Center.

Interest in embryo cryopreservation will be discussed with candidates before the start of IVF treatment. Women meeting the inclusion criteria who show no interest in embryo cryopreservation and in obtaining supernumerary embryos will be allocated to the mild stimulation (group A) protocol. Alternatively, women interested in obtaining a high number of embryos for the purpose of cryopreservation will be allocated to the conventional stimulation (group B) protocol.

ELIGIBILITY:
Inclusion Criteria:

* Female patients between 18-40 years of age
* Antral follicle count exceeding 16 and/or AMH exceeding 3.5 ng/dl
* PCOS features as per Rotterdam criteria: 2 of 3 criteria: a. Ultrasound morphology; b. Oligo/amenorrhea; c. Hyperandrogenism (clinical or chemical).

Exclusion Criteria:

* Recurrent implantation failure
* Recurrent pregnancy loss
* Congenital uterine anomalies
* Untreated maternal medical conditions (Diabetes, thyroid disease…)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — For women with PCOS who are undergoing IVF
Enrollment: 154 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | more than 24 weeks of gestation
  Defined as number of viable fetuses above 24 weeks of gestation per number of embryos transferred

SECONDARY OUTCOMES:
Total number of gonadotropins | up to 2 weeks
Duration of stimulation | up to 2 weeks
total number of developing follicles | up to 2 weeks
Rate of GnRHa trigger of final follicle maturation, endometrial thickness and pattern. | up to 2 weeks
Fertilization rate | up to 1 week
Cleavage rate | up to 1 week
Number of transferred embryos | up to 1 week
Quality of transferred embryos | up to 1 week
  Embryo grading as assessed on day 3 or day 5 (day of transfer)
Number of supernumerary embryos suitable for cryopreservation | up to 1 week
Treatment emergent adverse effects | up to 2 weeks
  headaches, hot flushes, irritability, visual changes, injection site discomfort, abdominal discomfort, and clinically significant OHSS (moderate and severe)
Cost | up to 2 weeks
  Direct and indirect costs of treatment will be recorded (ovarian stimulation agents, luteal support medications, OPU, ET, physician fees, monitoring)

CONTACTS AND LOCATIONS:
Overall Officials: Johnny T Awwad, M.D, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No